CLINICAL TRIAL: NCT03173638
Title: Phase II Safety Assessment of Intravitreal Injection of Mesenchymal Stem Cells for Acute Non Arteritic Anterior Ischemic Optic Neuropathy (NAION)
Brief Title: Safety Assessment of Intravitreal Mesenchymal Stem Cells for Acute Non Arteritic Anterior Ischemic Optic Neuropathy
Acronym: NEUROSTEM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: University of Valladolid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOBA01-2016; 2016-003029-40 (EudraCT Number)
Record Dates: First submitted 2017-05-24; First posted 2017-06-02 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Non Arteritic Ischemic Optic Neuropathy
Keywords: acute non arteritic anterior ischemic optic neuropathy; mesenchymal stem cells; intravitreal injection; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal stem from valladolid (MSV) (Experimental): Allogenic mesenchymal stem cells from bone marrow
  Interventions: Procedure: intravitreal injection of MSV

INTERVENTIONS:
Procedure: intravitreal injection of MSV — A unique intravitreal injection of MSV in acute fase of NAION

SUMMARY:
In this study the investigators propose to perform a Phase II Clinical Trial which seeks to evaluate the safety of cell therapy as a new treatment for patients who suffer from acute non-arteritic anterior ischemic optic neuropathy (NAION). If it is successful, a later study to assess efficacy will be performed.

This disease has an age-adjusted incidence rate of 10/100.000, and in many cases it results in blindness. Currently, there is no available treatment and second eye involvement occurs in approximately 15-25% of the cases.

All this background originates a particularly dramatic outcome for the patient. Therefore, it seems justified to evaluate new therapies that maintain or improve the visual function in these patients.

The Project includes a clinical trial whose purpose is the assessment of the safety of intravitreal administration of allogenic mesenchymal stem cells (MSC) in patients with NAION, a product in clinical research phase (PEI No. 15-007) already approved for other human clinical applications (PEI No. 15-007).

It can be considered that the therapy with intravitreal injection of MSC is a treatment option in patients with acute NAION, since through the paracrine properties of these cells (secretion of neurotrophic, immunomodulatory and anti-apoptotic factors) it may prevent or reduce the progression of axonal degeneration caused by this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute unilateral NAION (within two weeks after the first symptoms) with at least two of the following:

  1. Sudden and unpainful monocular vision loss
  2. Visual field defects
  3. Dyschromatopsia.
  4. Ocular nerve head edema.
  5. Afferent relative pupil defect.
* Patients ≥ 50 years old, able to freely give informed consent.
* Best corrected visual acuity (BCVA) ≤ 0,1 in study eye.
* Pseudophakia in study eye.
* Preserved pupil sphincter muscle motility
* Signed informed consent form before any study procedure.
* Signed data protection consent form before any study procedure.

Exclusion Criteria:

* Giant cell arteritis evidence (clinical history, Erythrocyte sedimentation rate (ESR), C-Reactive Protein)
* Evidence of any other etiology that may justify the optic neuropathy (even in the non-study eye)
* History of systemic vasculitis, multiple sclerosis, collagenopathies or previous cancer treatments.
* Hypersensitivity or allergy to any compound used in the study, including investigational medicinal product (IMP).
* Positive pregnancy test at baseline
* Participation in any other research study within 2 months

Ophthalmic exclusion criteria

* History of uveitis or active ocular inflammation
* History or evidence of glaucoma or high intraocular pressure ( ≥ 24 mmHg in either eye).
* Mean opacities or retinal pathologies in the study eye.
* Any previous vitreous or glaucoma surgery in the study eye
* Cataract surgery within 3 months in the study eye

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Absence of inflammatory reaction - Slit lamp exploration - SUN (Standardization of Uveitis Nomenclature) scale | Changes compared to baseline in visits V1 (1day), V2 (1week), V3 (1 month), V4 (3 months), V5 (6 months) and V6 (12months) and in any unscheduled visit any patient might need
  Following the SUN scale, the parameters that will be taken into account in the slit lamp exploration will be: cells and flare in anterior chamber, and vitreous flare

SECONDARY OUTCOMES:
Adverse events procedure-related (intravitreal injection) | Throughout the study after treatment in visits V1 (1day), V2 (1week), V3 (1 month), V4 (3 months), V5 (6 months) and V6 (12months) and in any unscheduled visit any patient might need
  Conjunctival haemorrhages, anterior chamber inflammation, changes in intraocular pressure, infectious endophthalmitis, vitreous inflammation, retinal detachment, choroidal detachment, corneal opacities, lens opacities, neovascularization, macular edema or any other adverse event that may appear

CONTACTS AND LOCATIONS:
Overall Officials: José C Pastor Jimeno, MD, PhD, Principal Investigator — IOBA-UVA
Locations (1):
- IOBA - Applied Ophthalmobiology Institute, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pastor JC, Pastor-Idoate S, Lopez-Paniagua M, Para M, Blazquez F, Murgui E, Garcia V, Coco-Martin RM. Intravitreal allogeneic mesenchymal stem cells: a non-randomized phase II clinical trial for acute non-arteritic optic neuropathy. Stem Cell Res Ther. 2023 Sep 21;14(1):261. doi: 10.1186/s13287-023-03500-7. PMID 37735668
- See also: European Union Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-003029-40/ES